CLINICAL TRIAL: NCT05917938
Title: Investigation of Pharmacokinetics, Safety and Tolerability of a Single Subcutaneous Dose of NNC0194-0499 in Participants With Various Degrees of Hepatic Impairment and Normal Hepatic Function
Brief Title: A Research Study Looking at How a Single Dose of the Study Medicine NNC0194-0499 Behaves in Participants With Reduced Liver Function Compared to Participants With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9500-4621; 2022-001835-10 (EudraCT Number); U1111-1278-1745 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-06-08; First posted 2023-06-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Impairment; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants With Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single subcutaneous dose of 30 milligram (mg) of NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499
- Participants With Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child Pugh Grade A) will receive a single subcutaneous dose of 30 mg of NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499
- Participants With Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Grade B) will receive a single subcutaneous dose of 30 mg of NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499
- Participants With Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh Grade C) will receive a single subcutaneous dose of 30 mg of NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499

INTERVENTIONS:
Drug: NNC0194-0499 — NNC0194-0499 will be administered subcutaneously in a skinfold in the thigh in the form of a solution for injection.

SUMMARY:
The study medicine NNC0194-0499 is under development for non-alcoholic fatty liver disease (NAFLD) including non-alcoholic steatohepatitis (NASH). All participants will receive a single dose of 30 milligram (mg) of the study medicine. The study medicine will be given in the form of an injection of 0.6 millilitres in a skinfold of the thigh (subcutaneous). The study will last for up to 64 days. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period. Women who are able to become pregnant must use highly effective contraception and will be counselled on the use of contraception. Participants with impaired liver function will undergo an ultrasound of the belly and measurement of brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-80 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.5-39.9 kilogram per square meter (kg/m^2) (both inclusive). Specific inclusion criterion only for participants with hepatic impairment:
* Participants with stable hepatic impairment classified as Child-Pugh grade A, B or C as assessed by the investigator. Stable hepatic impairment is defined as no clinically significant change in disease status, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
AUC0-∞, Single Dose, NNC0194-0499: the area under the NNC0194-0499 serum concentration-time curve from time 0 to infinity after a single dose | From 0 hours (Day 1) until end of study visit (Day 36)
  Measured in nanomoles hour per liter (nmol h/L).

SECONDARY OUTCOMES:
Cmax, NNC0194-0499: the maximum concentration of NNC0194-0499 in serum | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in nanomoles per liter (nmol/L).
tmax, NNC0194-0499: the time from dose administration to maximum serum concentration of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in hours.
t1/2, NNC0194-0499: the terminal half-life of NNC0194-0499 in serum | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in hours.
CL/F, NNC0194-0499: the apparent total serum clearance of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in liters per hour.
Vz/F, NNC0194-0499: apparent volume of distribution of NNC0194-0499 after a single dose | From Day 1 (pre-dose) until completion of the end of trial visit (Day 36)
  Measured in liters.
Number of treatment emergent adverse events (TEAEs) | From time of trial product administration (Visit 2, Day 1) until completion of the end of trial visit (Visit 8, Day 36)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (5):
- APEX Research, München, Germany
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - Cardiomedicum Sp. z o.o., Krakow
- Slovakia (2):
  - Summit Clinical Research s.r.o., Bratislava
  - Summit Clinical Research s.r.o., Malacky

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com